CLINICAL TRIAL: NCT00188591
Title: Pilot Study to Investigate the Feasibility of Optical Spectroscopy to Quantify Bulk Breast Tissue Properties in Girls Age 10 - 14 Years
Brief Title: Light Based Analysis of Developing Breast Tissue in Adolescent Girls: a Feasibility Study
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Lothar Lilge, University Health Network
Other Study IDs: UHNREB#05-0154-CE; HC#92740
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Breast Cancer
Keywords: Optical Transillumination Spectroscopy; Breast Cancer Risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed pilot study attempts to investigate the feasibility of Optical Spectroscopy (OS) as a method to quantify breast tissue composition and density in adolescent females. Our goals include: to assess whether adolescent girls can be instructed to assist with the OS measurement procedure and to determine the OS technique's ability to show breast tissue composition and density in adolescent breast tissue.

DETAILED DESCRIPTION:
The period between menarche and the age of first full-term pregnancy has been identified as being most crucial for establishing an individual's future breast cancer risk. Epidemiological studies further suggest exposures, such as foods and toxins, during adolescence to have a significant impact on the likelihood of transformation in the developing breast resulting in cancer later in life. Adolescent diet affects mammary development directly and indirectly by influencing the micronutrients and the hormonal status of the adolescent. The goal of this study is to investigate the feasibility of Optical Spectroscopy (OS), a method based on differential light scattering and absorption in tissue, to quantify bulk breast tissue properties in adolescent females.

ELIGIBILITY:
Inclusion Criteria (Girls):

* Are in good health and are able to provide assent
* Are between the ages of 10 and 14
* Are interested in participating in this study
* Are willing to come, accompanied by a parent, to the Princess Margaret Hospital

Inclusion Criteria (Parents):

* Are able to provide consent
* Are willing to accompany your daughter to the Princess Margaret Hospital for one visit of about 45 minutes

Exclusion Criteria (Girls):

* Have had previous surgeries to the chest area

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Residents of Toronto, Ontario, Canada.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2005-04; Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Lilge, PhD, Principal Investigator — Ontario Cancer Institute, University Health Network, Toronto, Ontario, Canada M5G 2M9; Department of Biophysics and Bioimaging, University of Toronto, Toronto, Ontario, Canada M5G 2M9
Locations (1):
- University Health Network / Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Blyschak K, Simick M, Jong R, Lilge L. Classification of breast tissue density by optical transillumination spectroscopy: optical and physiological effects governing predictive value. Med Phys. 2004 Jun;31(6):1398-414. doi: 10.1118/1.1738191. PMID 15259643
- [Background] Simick MK, Jong R, Wilson B, Lilge L. Non-ionizing near-infrared radiation transillumination spectroscopy for breast tissue density and assessment of breast cancer risk. J Biomed Opt. 2004 Jul-Aug;9(4):794-803. doi: 10.1117/1.1758269. PMID 15250768
- [Background] Blackmore KM, Knight JA, Jong R, Lilge L. Assessing breast tissue density by transillumination breast spectroscopy (TIBS): an intermediate indicator of cancer risk. Br J Radiol. 2007 Jul;80(955):545-56. doi: 10.1259/bjr/26858614. Epub 2007 May 30. PMID 17537757
- [Background] Simick MK, Lilge L. Optical transillumination spectroscopy to quantify parenchymal tissue density: an indicator for breast cancer risk. Br J Radiol. 2005 Nov;78(935):1009-17. doi: 10.1259/bjr/14696165. PMID 16249602